CLINICAL TRIAL: NCT05124483
Title: Anti-COVID19 VaccinaTion AKS-452 BOOSTER (ACT-BOOSTER Study)
Acronym: ACT-BOOSTER
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medical Center Groningen (Other)
Collaborators: TRACER Europe BV (Industry); PRA Health Sciences (Industry)
Responsible Party: Principal Investigator, Schelto Kruijff, MD PhD, prof dr, University Medical Center Groningen
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 900452-CT-21-001
Record Dates: First submitted 2021-11-17; First posted 2021-11-18 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: COVID-19
Keywords: COVID-19; Vaccine; Booster
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Single center, open-label, safety and efficacy study on the biological activity of a SP/RBD-Fc antigen booster vaccine (AKS-452X) against COVID-19.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Pfizer [Comirnaty] (Experimental): To determine the immunogenicity 4-6 weeks after subcutaneous injection of a booster dose of 90 µg AKS-452X vaccine given at >=3 months post-initial vaccination with the registered Pfizer [Comirnaty] vaccine.
  Interventions: Biological: AKS-452X
- Moderna [Spikevax] (Experimental): To determine the immunogenicity 4-6 weeks after subcutaneous injection of a booster dose of 90 µg AKS-452X vaccine given at >=3 months post-initial vaccination with the registered Moderna [Spikevax] vaccine.
  Interventions: Biological: AKS-452X
- Janssen [Ad26.COV2.S] (Experimental): To determine the immunogenicity 4-6 weeks after subcutaneous injection of a booster dose of 90 µg AKS-452X vaccine given at >=3 months post-initial vaccination with the registered Janssen [Ad26.COV2.S] vaccine.
  Interventions: Biological: AKS-452X
- AstraZeneca [Vaxzevria]) (Experimental): To determine the immunogenicity 4-6 weeks after subcutaneous injection of a booster dose of 90 µg AKS-452X vaccine given at >=3 months post-initial vaccination with the registered AstraZeneca [Vaxzevria]) vaccine.
  Interventions: Biological: AKS-452X

INTERVENTIONS:
Biological: AKS-452X — subcutaneous injection of 90 µg AKS-452X

SUMMARY:
Aim: To investigate if a subcutaneous (s.c.) booster dose of 90 µg of the naked Akston AKS-452 vaccine (AKS-452X) at >= 3 months post initial vaccination, with any of the four registered vaccines, will boost the antibody titer and immune response in human healthy volunteers 4-6 weeks after s.c. injection.

DETAILED DESCRIPTION:
Hypothesis: A booster dose of naked (i.e. non-adjuvanted) AKS-452 vaccine will provide an enhanced immune response after vaccination with any of the registered vaccines against COVID-19.

Primary objective: To determine the immunogenicity 4-6 weeks after subcutaneous injection of a booster dose of AKS-452X vaccine given at >=3 months post-initial vaccination (i.e. Pfizer [ Comirnaty], Moderna [Spikevax], Janssen [Ad26.COV2.S], AstraZeneca [Vaxzevria]) in human healthy volunteers.

Secondary objective: Vaccine safety and side effects after booster vaccination. Follow-up will occur for up to 9 months post-study vaccine.

Study design: Single center, open-label, safety and efficacy study on the biological activity of a SP/RBD-Fc antigen booster vaccine (AKS-452X) against COVID-19.

Study population: Healthy human volunteers, 18 - 85 years, having received a registered vaccine (i.e. Pfizer [Comirnaty], Moderna [Spikevax], Janssen [Ad26.COV2.S], AstraZeneca [Vaxzevria]).

Intervention: One booster dose-level of naked AKS-452 (90 µg) administered via s.c. route in 150 subjects per cohort in which safety parameters and neutralizing IgG titers will be reviewed after the booster dose of 90 µg s.c.. Enhanced immune response is defined as: i) seroconversion based on a true positive based on the SP/RBD IgG ELISA assay positive/negative cutoff criteria using the quantitative cut-off value defined by the assay kit batch expressed in μg/mL. The positive/negative cutoff value was established as 2.42 µg/mL from the validation analysis for the current lot of assay kits, but it should be noted that for each new lot of assay kits, Akston QC performs a re-validation of the cutoff value in order to maintain clinical agreement from lot-to-lot, ii) two times (2x) the baseline SP/RBD IgG at day 56 after a boostering, as compared to the titer at the time of screening.

Main study parameters/endpoints: Primary endpoint: The percentage of patients that i) achieve an SP/RBD-specific IgG antibody titer level of ≥ 2.42 µg/mL at the day 28 time-point post-intervention (i.e. booster vaccine) if the base-line value prior to receiving the booster vaccine was < 2.42 µg/mL or ii) where the SP/RBD-specific IgG antibody titer is at least 2x the base-line value prior to receiving the booster vaccine if the base-line value prior to receiving the booster vaccine was ≥ 2.42 µg/mL. The percentage of patients in each of the four cohorts that achieve the primary endpoint threshold at 28 days post-intervention will be calculated (n (%)). Secondary endpoint: Safety evaluation in the four cohorts for local and systemic adverse events after injection at each pre-defined scheduled follow-up (at 28, 56, 91, 182 and 238 days post intervention). Patients will continue to be followed passively for additional safety events out to 9 months post-intervention.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, a subject must meet all of the following criteria:

* Age 18-85 years (extremes included), males and females.
* Negative SARS-CoV-2 serology (an anti-SARS-CoV-2 SP-specific IgG ELISA)
* Body mass index (BMI) between 19.0 and 30.0 kg/m2, inclusive
* General good health, without significant medical illness, as determined via physical exam findings, or vital signs
* No clinically significant laboratory abnormalities as determined by the investigator

  o Note: one retest of lab tests is allowed within the screening window
* Informed Consent Form signed voluntarily before any study-related procedure is performed, indicating that the subject understands the purpose and procedures required for the study and is willing to participate in the study
* Willing to adhere to the prohibitions and restrictions specified in this protocol
* All participants have received a completed (registered) vaccine at least 3 months before inclusion in this study (i.e. Pfizer [Comirnaty], Moderna [Spikevax], Janssen [Ad26.COV2.S], AstraZeneca [Vaxzevria]).
* Negative hepatitis panel (including hepatitis B surface Ag and anti-hepatitis C virus Abs) and negative human immunodeficiency virus Ab and Ag screens at screening
* Female subjects should fulfil one of the following criteria:

  * At least 1 year post-menopausal (amenorrhea >12 months
  * Surgically sterile (bilateral oophorectomy, hysterectomy, or tubal ligation);
  * Will use adequate forms of contraceptives from screening to discharge.
* Female subjects of childbearing potential and male subjects who are sexually active with a female partner of childbearing potential must agree to the use of an effective method of birth control from screening to discharge

  o Note: medically acceptable methods of contraception that may be used by the subject and/or partner include combined oral contraceptive, contraceptive vaginal ring, contraceptive injection, intrauterine device, etonogestrel implant, double barrier, sterilization and vasectomy
* Female subject has a negative pregnancy test at screening and upon check-in at the clinical site.

  * Note: pregnancy testing will consist of a serum pregnancy test at screening and urine pregnancy tests at the dosing visit, in all women.

Exclusion Criteria:

* Pregnant or breast-feeding females
* Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, hematologic, rheumatologic, endocrine, autoimmune, or renal disease
* Any laboratory test which is abnormal, and which is deemed by the Investigator(s) to be clinically significant
* Behavioral or cognitive impairment or psychiatric disease that in the opinion of the investigator affects the ability of the subject to understand and cooperate with the study protocol
* Current alcohol/illicit drug/nicotine abuse or addiction: history or evidence of current drug use or addiction (positive drug screen for amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, or opiates) or signs of excessive use of alcohol at screening and at day 0.
* Presence of any febrile illness (T > = 38.0°C or lab confirmed viral disease (PCR)) or symptoms suggestive of a viral respiratory infection within 1 weeks prior to vaccination. Participants will be screened for SARS-Cov-2 with an EUA-approved PCR test at screening, and at day 0.
* Use of corticosteroids (excluding topical preparations for cutaneous or nasal use) or use of immunosuppressive drugs within 30 days before inoculation
* A history of anaphylaxis, history of allergic reaction to vaccine, known allergy to one of the components in AKS-452X. Mild allergies without angio-edema or treatment need can be included if deemed not to be of clinical significance (including but not limited to allergy to animals or mild seasonal hay fever)
* A history of asthma within the past 10 years, or a current diagnosis of asthma or reactive airway disease associated with exercise
* Receipt of blood or blood-derived products (including immunoglobulin) within 6 months prior to vaccination.
* Receipt of another investigational agent within 30 days or 5 times the product half-life (whichever is longest) prior to vaccination
* Deprived of freedom by an administrative or court order or in an emergency setting
* Any condition that in the opinion of the principal investigator (PI) would jeopardize the safety or rights of a person participating in the trial or would render the person unable to comply with the protocol.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2022-04-21 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
Enhanced Immune Response | 28 days post-injection of the booster AKS-452X
  The percentage of patients that i) achieve an SP/RBD-specific IgG antibody titer level of ≥ 2.42 µg/mL at the day 28 time-point post-intervention (i.e. booster vaccine) if the base-line value prior to receiving the booster vaccine was < 2.42 µg/mL or ii) where the SP/RBD-specific IgG antibody titer is at least 2x the base-line value prior to receiving the booster vaccine if the base-line value prior to receiving the booster vaccine was ≥ 2.42 µg/mL. The percentage of patients in each of the four cohorts that achieve the primary endpoint threshold at 28 days post-intervention will be calculated (n (%)).

SECONDARY OUTCOMES:
Safety evaluation | 9 months post-injection of the booster AKS-452X
  Safety evaluation in the four cohorts for local and systemic adverse events after injection at each pre-defined scheduled follow-up (at 28, 56, 91, 182 and 238 days post intervention). Patients will continue to be followed passively for additional safety events out to 9 months post-intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Gooitzen M van Dam, MD, PhD, Study Chair — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No